CLINICAL TRIAL: NCT03002766
Title: Ten Years Results of a Score System to Address Adjuvant Therapies After Breast Conserving Surgery for Ductal Carcinoma in Situ of the Breast.
Acronym: DCIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 67/13
Record Dates: First submitted 2016-12-02; First posted 2016-12-26 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Carcinoma Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Breast conservative surgery

SUMMARY:
By this non-randomized prospective study, it's evaluated the outcome of patients underwent BCS for DCIS at whom an established score system to address adjuvant therapies have been prospectively applied, according to the wideness of free margins.

Between March 2000 and April 2006, 224 patients were enrolled and followed within the study.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years;
* female candidate to breast conservative surgery

Exclusion Criteria:

* female with previous omolateral or controlateral breast cancer;
* female with previous radiotherapy (RT).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2000-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Ipsilateral Breast Tumor Recurrence (IBTR) | six years

SECONDARY OUTCOMES:
Contralateral breast cancer (CBC) | six years
  the side effects of radiotherapy may outweigh the reduction in the risk of IBTR

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Gennaro, MD, Principal Investigator — Fondazione IRCCS ISTITUTO NAZIONALE TUMORI
Locations (1):
- Massimiliano Gennaro, Milan, MI, Italy

REFERENCES:
- [Background] Kaplan EL, Meier P. Nonparametric estimation from incomplete observations. J AM Stat Assoc 53:457-481, 1958.
- [Result] Fisher B, Dignam J, Wolmark N, Mamounas E, Costantino J, Poller W, Fisher ER, Wickerham DL, Deutsch M, Margolese R, Dimitrov N, Kavanah M. Lumpectomy and radiation therapy for the treatment of intraductal breast cancer: findings from National Surgical Adjuvant Breast and Bowel Project B-17. J Clin Oncol. 1998 Feb;16(2):441-52. doi: 10.1200/JCO.1998.16.2.441. PMID 9469327
- [Result] Donker M, Litiere S, Werutsky G, Julien JP, Fentiman IS, Agresti R, Rouanet P, de Lara CT, Bartelink H, Duez N, Rutgers EJ, Bijker N. Breast-conserving treatment with or without radiotherapy in ductal carcinoma In Situ: 15-year recurrence rates and outcome after a recurrence, from the EORTC 10853 randomized phase III trial. J Clin Oncol. 2013 Nov 10;31(32):4054-9. doi: 10.1200/JCO.2013.49.5077. Epub 2013 Sep 16. PMID 24043739
- [Result] Holmberg L, Garmo H, Granstrand B, Ringberg A, Arnesson LG, Sandelin K, Karlsson P, Anderson H, Emdin S. Absolute risk reductions for local recurrence after postoperative radiotherapy after sector resection for ductal carcinoma in situ of the breast. J Clin Oncol. 2008 Mar 10;26(8):1247-52. doi: 10.1200/JCO.2007.12.7969. Epub 2008 Feb 4. PMID 18250350
- [Result] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Correa C, McGale P, Taylor C, Wang Y, Clarke M, Davies C, Peto R, Bijker N, Solin L, Darby S. Overview of the randomized trials of radiotherapy in ductal carcinoma in situ of the breast. J Natl Cancer Inst Monogr. 2010;2010(41):162-77. doi: 10.1093/jncimonographs/lgq039. PMID 20956824
- [Result] Cuzick J, Sestak I, Pinder SE, Ellis IO, Forsyth S, Bundred NJ, Forbes JF, Bishop H, Fentiman IS, George WD. Effect of tamoxifen and radiotherapy in women with locally excised ductal carcinoma in situ: long-term results from the UK/ANZ DCIS trial. Lancet Oncol. 2011 Jan;12(1):21-9. doi: 10.1016/S1470-2045(10)70266-7. Epub 2010 Dec 7. PMID 21145284
- [Result] Fisher B, Dignam J, Wolmark N, Wickerham DL, Fisher ER, Mamounas E, Smith R, Begovic M, Dimitrov NV, Margolese RG, Kardinal CG, Kavanah MT, Fehrenbacher L, Oishi RH. Tamoxifen in treatment of intraductal breast cancer: National Surgical Adjuvant Breast and Bowel Project B-24 randomised controlled trial. Lancet. 1999 Jun 12;353(9169):1993-2000. doi: 10.1016/S0140-6736(99)05036-9. PMID 10376613
- [Result] Margolese RG, Cecchini RS, Julian TB, Ganz PA, Costantino JP, Vallow LA, Albain KS, Whitworth PW, Cianfrocca ME, Brufsky AM, Gross HM, Soori GS, Hopkins JO, Fehrenbacher L, Sturtz K, Wozniak TF, Seay TE, Mamounas EP, Wolmark N. Anastrozole versus tamoxifen in postmenopausal women with ductal carcinoma in situ undergoing lumpectomy plus radiotherapy (NSABP B-35): a randomised, double-blind, phase 3 clinical trial. Lancet. 2016 Feb 27;387(10021):849-56. doi: 10.1016/S0140-6736(15)01168-X. Epub 2015 Dec 11. PMID 26686957
- [Result] Forbes JF, Sestak I, Howell A, Bonanni B, Bundred N, Levy C, von Minckwitz G, Eiermann W, Neven P, Stierer M, Holcombe C, Coleman RE, Jones L, Ellis I, Cuzick J; IBIS-II investigators. Anastrozole versus tamoxifen for the prevention of locoregional and contralateral breast cancer in postmenopausal women with locally excised ductal carcinoma in situ (IBIS-II DCIS): a double-blind, randomised controlled trial. Lancet. 2016 Feb 27;387(10021):866-73. doi: 10.1016/S0140-6736(15)01129-0. Epub 2015 Dec 11. PMID 26686313
- [Result] Povoski SP, Jimenez RE, Wang WP, Xu RX. Standardized and reproducible methodology for the comprehensive and systematic assessment of surgical resection margins during breast-conserving surgery for invasive breast cancer. BMC Cancer. 2009 Jul 27;9:254. doi: 10.1186/1471-2407-9-254. PMID 19635166
- [Result] Rizzo M, Iyengar R, Gabram SG, Park J, Birdsong G, Chandler KL, Mosunjac MB. The effects of additional tumor cavity sampling at the time of breast-conserving surgery on final margin status, volume of resection, and pathologist workload. Ann Surg Oncol. 2010 Jan;17(1):228-34. doi: 10.1245/s10434-009-0643-x. Epub 2009 Jul 28. PMID 19636625
- [Result] Mantel N. Evaluation of survival data and two new rank order statistics arising in its consideration. Cancer Chemother Rep. 1966 Mar;50(3):163-70. No abstract available. PMID 5910392
- [Result] EORTC Breast Cancer Cooperative Group; EORTC Radiotherapy Group; Bijker N, Meijnen P, Peterse JL, Bogaerts J, Van Hoorebeeck I, Julien JP, Gennaro M, Rouanet P, Avril A, Fentiman IS, Bartelink H, Rutgers EJ. Breast-conserving treatment with or without radiotherapy in ductal carcinoma-in-situ: ten-year results of European Organisation for Research and Treatment of Cancer randomized phase III trial 10853--a study by the EORTC Breast Cancer Cooperative Group and EORTC Radiotherapy Group. J Clin Oncol. 2006 Jul 20;24(21):3381-7. doi: 10.1200/JCO.2006.06.1366. Epub 2006 Jun 26. PMID 16801628
- [Result] Rutgers EJ; EUSOMA Consensus Group. Quality control in the locoregional treatment of breast cancer. Eur J Cancer. 2001 Mar;37(4):447-53. doi: 10.1016/s0959-8049(00)00386-5. No abstract available. PMID 11267852
- [Result] Schwartz GF, Veronesi U, Clough KB, Dixon JM, Fentiman IS, Heywang-Kobrunner SH, Holland R, Hughes KS, Mansel RE, Margolese R, Mendelson EB, Olivotto IA, Palazzo JP, Solin LJ; Consensus Conference Committee. Consensus conference on breast conservation. J Am Coll Surg. 2006 Aug;203(2):198-207. doi: 10.1016/j.jamcollsurg.2006.04.009. No abstract available. PMID 16864033
- [Result] Rutqvist LE, Rose C, Cavallin-Stahl E. A systematic overview of radiation therapy effects in breast cancer. Acta Oncol. 2003;42(5-6):532-45. doi: 10.1080/02841860310014444. PMID 14596511
- [Result] Healy C, Allen RJ Sr. The evolution of perforator flap breast reconstruction: twenty years after the first DIEP flap. J Reconstr Microsurg. 2014 Feb;30(2):121-5. doi: 10.1055/s-0033-1357272. Epub 2013 Oct 25. PMID 24163223
- [Result] Kasem A, Wazir U, Headon H, Mokbel K. Breast lipofilling: a review of current practice. Arch Plast Surg. 2015 Mar;42(2):126-30. doi: 10.5999/aps.2015.42.2.126. Epub 2015 Mar 16. PMID 25798382
- [Result] Gennaro M, Ferraris C, Guida V, Tomasic G, Carcangiu ML, Greco M. Conservative surgery in breast cancer. Significance of resection margins. Breast. 2001 Oct;10(5):432-7. doi: 10.1054/brst.2001.0297. PMID 14965620
- [Result] Macdonald HR, Silverstein MJ, Lee LA, Ye W, Sanghavi P, Holmes DR, Silberman H, Lagios M. Margin width as the sole determinant of local recurrence after breast conservation in patients with ductal carcinoma in situ of the breast. Am J Surg. 2006 Oct;192(4):420-2. doi: 10.1016/j.amjsurg.2006.06.031. PMID 16978941
- [Result] Van Zee KJ, Liberman L, Samli B, Tran KN, McCormick B, Petrek JA, Rosen PP, Borgen PI. Long term follow-up of women with ductal carcinoma in situ treated with breast-conserving surgery: the effect of age. Cancer. 1999 Nov 1;86(9):1757-67. doi: 10.1002/(sici)1097-0142(19991101)86:93.0.co;2-v. PMID 10547549
- [Result] Fisher ER, Dignam J, Tan-Chiu E, Costantino J, Fisher B, Paik S, Wolmark N. Pathologic findings from the National Surgical Adjuvant Breast Project (NSABP) eight-year update of Protocol B-17: intraductal carcinoma. Cancer. 1999 Aug 1;86(3):429-38. doi: 10.1002/(sici)1097-0142(19990801)86:33.0.co;2-y. PMID 10430251
- [Result] Simpson PT, Reis-Filho JS, Lambros MB, Jones C, Steele D, Mackay A, Iravani M, Fenwick K, Dexter T, Jones A, Reid L, Da Silva L, Shin SJ, Hardisson D, Ashworth A, Schmitt FC, Palacios J, Lakhani SR. Molecular profiling pleomorphic lobular carcinomas of the breast: evidence for a common molecular genetic pathway with classic lobular carcinomas. J Pathol. 2008 Jul;215(3):231-44. doi: 10.1002/path.2358. PMID 18473330
- [Result] Lesurf R, Aure MR, Mork HH, Vitelli V; Oslo Breast Cancer Research Consortium (OSBREAC); Lundgren S, Borresen-Dale AL, Kristensen V, Warnberg F, Hallett M, Sorlie T. Molecular Features of Subtype-Specific Progression from Ductal Carcinoma In Situ to Invasive Breast Cancer. Cell Rep. 2016 Jul 26;16(4):1166-1179. doi: 10.1016/j.celrep.2016.06.051. Epub 2016 Jul 7. PMID 27396337
- [Result] Silverstein MJ, Lagios MD, Craig PH, Waisman JR, Lewinsky BS, Colburn WJ, Poller DN. A prognostic index for ductal carcinoma in situ of the breast. Cancer. 1996 Jun 1;77(11):2267-74. doi: 10.1002/(SICI)1097-0142(19960601)77:113.0.CO;2-V. PMID 8635094
- [Result] Silverstein MJ, Lagios MD. Treatment selection for patients with ductal carcinoma in situ (DCIS) of the breast using the University of Southern California/Van Nuys (USC/VNPI) prognostic index. Breast J. 2015 Mar-Apr;21(2):127-32. doi: 10.1111/tbj.12368. Epub 2015 Jan 20. PMID 25600630
- [Result] Sagara Y, Freedman RA, Vaz-Luis I, Mallory MA, Wong SM, Aydogan F, DeSantis S, Barry WT, Golshan M. Patient Prognostic Score and Associations With Survival Improvement Offered by Radiotherapy After Breast-Conserving Surgery for Ductal Carcinoma In Situ: A Population-Based Longitudinal Cohort Study. J Clin Oncol. 2016 Apr 10;34(11):1190-6. doi: 10.1200/JCO.2015.65.1869. Epub 2016 Feb 1. PMID 26834064
- [Result] Benson JR, Jatoi I, Toi M. Treatment of low-risk ductal carcinoma in situ: is nothing better than something? Lancet Oncol. 2016 Oct;17(10):e442-e451. doi: 10.1016/S1470-2045(16)30367-9. PMID 27733270